CLINICAL TRIAL: NCT04940923
Title: Does Peripheral Neuroinflammation Predict Chronicity Following Whiplash?
Brief Title: Neuroinflammation as a Predictor of Chronicity in Whiplash
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sussex (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 278291/ 070 DIL
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Whiplash Injuries
Keywords: Magnetic resonance imaging; Pain threshold; Neuritis; Prognosis
MeSH Terms: conditions — Whiplash Injuries; Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients within 4 weeks of a whiplash injury.
  Interventions: Diagnostic Test: MRI
- Healthy controls: Age and gender matched healthy controls
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — T2 weighted and DTI MRI images of brachial plexus and wrist. Quantitative sensory tests include warm and cold detection and pain thresholds, paradoxical heat sensation, mechanical detection thresholds, mechanical pain sensation and thresholds, wind up ratios, vibration thresholds and pressure pain thresholds.
  Clinical tests include standard neurological tests and test for heightened nerve mechanosensitivity.
  Blood serum to analyse inflammatory proteins. Questionnaires include neck disability index, painDETECT, PTSD8, pain catastrophising scale, eq-5D-5L, DASS 42 and global perceived recovery
  Other Names: Quantitative sensory tests; Blood serum tests; Clinical tests; Questionnaires

SUMMARY:
Whiplash describes an injury to the neck caused by a rapid movement of the head. It often occurs during a motor vehicle collision, causing considerable pain and distress. Most patients are diagnosed with whiplash associated disorder grade-2 (WAD2). Half of these patients develop chronic pain. Current treatments for patients are ineffective. It is difficult to predict which patients will develop chronic pain, and therefore how to manage these patients. The characteristics of pain felt by many patients with WAD2 suggests that symptoms are caused by an injury to the nerves in the neck and arm. However, on clinical examination there is no indication that these nerves are significantly injured.

Work from the investigators' laboratory suggests that nerves may be inflamed. In this study, the contribution of nerve inflammation to symptoms early following whiplash will be established. It will determine whether clinical tests are able to identify those patients with inflamed nerves. It will also determine whether the presence of nerve inflammation can be used to identify patients who develop chronic pain. The study will recruit 115 patients within one month following a whiplash injury and thirty-two healthy volunteers. Participants will undergo a clinical assessment. A blood sample will be taken to look for inflammatory proteins and magnetic resonance imaging will be used to identify nerve inflammation in the neck and wrist. Questionnaires to establish neck disability, pain quality and psychological distress will be completed. MRI findings will be compared to healthy controls. At six-months, patients will be asked to repeat the questionnaires, which will be used to identify those patients who have recovered. Twenty-five recovered and twenty-five non-recovered patients will undergo a repeat MRI and clinical assessment. Although patients on this study will not directly benefit, the findings will help with early diagnosis and could refocus treatment to reduce chronic pain.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Male and female patients with chronic whiplash associated disorder that meet the Quebec Task Force Classification of whiplash grade II
2. Within approximately four weeks of their whiplash injury
3. Age 18-60
4. Participants capable of giving informed consent

Healthy Volunteers:

1. Free of neck or upper limb pain
2. No history of a whiplash injury or of neck or arm pain lasting >3 months or any recent cervical or upper limb trauma requiring medical treatment.
3. Age 18-60
4. Participants capable of giving informed consent

Exclusion Criteria:

Patients:

1. Diagnosis of whiplash grade I (neck complaints without physical signs), III (obvious neurological signs) or IV (fracture or dislocation)
2. Experienced concussion or loss of consciousness as a result of the accident
3. Previous history of whiplash
4. Previous history of neck pain or headaches that required treatment

   All participants (patients and healthy volunteers):
5. Unsuitability to undergo MRI (assessed with the MRI screening questionnaire)
6. Pregnant
7. History of inflammatory disease (e.g. autoimmune diseases, rheumatoid arthritis), neuropathy, diabetes, cancer or non-medically controlled hypertension
8. Current ongoing steroid treatment
9. Participants with an inadequate understanding of English will also be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People who have sustained a whiplash injury less than 4 weeks prior to their participation in the study.
  Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
MRI T2-weighted nerve signal strength | Baseline
  T2-weighted nerve signal strength in the brachial plexus and median nerve compared to healthy control group
Change in MRI T2-weighted nerve signal strength | From baseline to 6 months
  Change in T2-weighted nerve signal strength in the brachial plexus and median nerve at 6 months compared to baseline
Fractional anisotropy from diffusion tensor images | Baseline
  Fractional anisotropy measurements from brachial plexus and median nerve compared to healthy controls
Change in fractional anisotropy from Diffusion tensor images | From baseline to 6 months
  Fractional anisotropy from brachial plexus and median nerve compared to baseline

SECONDARY OUTCOMES:
T1 MRI median nerve morphology | Baseline
  ratio/mm2; continuous data
Changes to T1 MRI median nerve morphology | From baseline to 6 months
  ratio/mm2; continuous data
Pro-inflammatory cytokine levels | Baseline
  Proinflammatory cytokine assay (pg/ml) continuous data
Change in Pro-inflammatory cytokine levels | From baseline to 6 months
  Proinflammatory cytokine assay (pg/ml) continuous data
Tests for heightened nerve mechanosensitivity- upper limb neurodynamic test (median nerve) | Baseline
  Measures heightened response to tensile load applied to the nerve. Range of elbow extension at point of symptoms (degrees)
Change to tests for heightened nerve mechanosensitivity- upper limb neurodynamic test (median nerve) | From baseline to 6 months
  Measures heightened response to tensile load applied to the nerve. Range of elbow extension at point of symptoms (degrees)
Tests for heightened nerve mechanosensitivity- Pressure pain threshold | Baseline
  Algometer applied to ulnar nerve at the cubital tunnel and median nerve at carpal tunnel. Pressure pain threshold (Kg) at point of change from pressure to pain.
Change in heightened nerve mechanosensitivity- Pressure pain threshold | From baseline to 6 months
  Algometer applied to ulnar nerve at the cubital tunnel and median nerve at carpal tunnel. Pressure pain threshold (Kg) at point of change from pressure to pain.
Quantitative sensory testing- warm and cold pain thresholds | Baseline
  Thresholds measured over index finger using a thermotester- continuous data measured in degrees Celsius (point at which the probe changes to warm pain or cold pain)
Change to Quantitative sensory testing- warm and cold pain thresholds | From baseline to 6 months
  Thresholds measured over index finger using a thermotester- continuous measured in degrees Celsius (point at which the probe changes to warm pain or cold pain)
Quantitative sensory testing- Mechanical pain threshold | Baseline
  Thresholds measured over index finger using a series of weighted pin prick stimulators (mN). Participant scores pain from 0-100 for each stimulus applied. Geometric mean calculated
Change in Quantitative sensory testing- Mechanical pain threshold | From baseline to 6 months
  Thresholds measured over index finger using a series of weighted pin prick stimulators (mN). Participant scores pain from 0-100 for each stimulus applied. Geometric mean calculated
Quantitative sensory testing- Pressure pain threshold | Baseline
  Thresholds measured over thenar eminance using an algometer (Kg). Pressure applied and participant indicates when pressure changes to pain (mean of 3)
Change in quantitative sensory testing- Pressure pain threshold | From baseline to 6 months
  Thresholds measured over thenar eminance using an algometer (Kg). Pressure applied and participant indicates when pressure changes to pain (mean of 3)
Changes in Pain levels on Visual analogue scale | From baseline to 6 months
  Participant indicated pain level on a 10cm scale of 0-10
Change in Neck disability index | From baseline to 6 months
  Neck disability index. Scale -10 questions each scored 0-5. Total score /50
Change in painDETECT questionnaire | From baseline to 6 months
  A measure of neuropathic pain. A continuous scale: 0-38 or trichotomised: no, unclear, yes. A score of >19 suggests neuropathic pain.
Change in Short post-traumatic stress inventory | From baseline to 6 months
  A measure of post traumatic stress - 8 questions scale of 0-3

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dilley, PhD, Principal Investigator — Brighton and Sussex Medical School
Locations (2):
- United Kingdom (2):
  - Brighton and Sussex Medical School, Brighton, East Sussex
  - Oxford Neuroscience, University of Oxford, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ridehalgh C, Fundaun J, Bremner S, Cercignani M, Koushesh S, Schmid AB, Dilley A. Temporal development of peripheral neuroinflammation in whiplash-associated disorder grade II and its role in chronicity. Pain. 2026 Feb 1;167(2):356-371. doi: 10.1097/j.pain.0000000000003816. Epub 2025 Oct 10. PMID 41081757
- [Derived] Ridehalgh C, Fundaun J, Bremner S, Cercignani M, Koushesh S, Young R, Novak A, Greening J, Schmid AB, Dilley A. Evidence for peripheral neuroinflammation after acute whiplash. Pain. 2025 Oct 1;166(10):2285-2299. doi: 10.1097/j.pain.0000000000003560. Epub 2025 Mar 4. PMID 40035629
- [Derived] Ridehalgh C, Fundaun J, Bremner S, Cercignani M, Young R, Trivedy C, Novak A, Greening J, Schmid A, Dilley A. Does peripheral neuroinflammation predict chronicity following whiplash injury? Protocol for a prospective cohort study. BMJ Open. 2022 Dec 15;12(12):e066021. doi: 10.1136/bmjopen-2022-066021. PMID 36521884